CLINICAL TRIAL: NCT02981082
Title: A Double-blinded, Placebo-controlled Pilot Study of Dimethyl Fumarate (DMF) in Pulmonary Arterial Hypertension (PAH) Associated With Systemic Sclerosis (SSc-PAH): The Effect of DMF on Clinical Disease and Biomarkers of Oxidative Stress.
Brief Title: Dimethyl Fumarate (DMF) in Systemic Sclerosis-Associated Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Robert Lafyatis (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, Robert Lafyatis, Professor of Medicine and the Thomas Medsger Professor in Arthritis Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO16070614
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Systemic Sclerosis; Pulmonary; Hypertension
Keywords: Systemic Sclerosis, Scleroderma, PAH, Pulmonary Hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary; Scleroderma, Diffuse | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dimethyl Fumarate (DMF) (Active Comparator): Twice daily oral doses of Dimethyl Fumarate (DMF) 120mg for the first 7 days followed by the maintenance dose of Dimethyl Fumarate (DMF) 240mg twice a day. Subjects will be dosed for 24 weeks
  Interventions: Drug: Dimethyl Fumarate (DMF)
- Placebo (Placebo Comparator): Twice daily oral doses of placebo for 12 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dimethyl Fumarate (DMF) — Dimethyl Fumarate (DMF) is a prescription medicine used to treat relapsing multiple sclerosis.
  Other Names: Tecfidera
  Arms: Dimethyl Fumarate (DMF)
Drug: Placebo Oral Tablet — Sugar pill manufactured to mimic Dimethyl Fumarate (DMF)
  Arms: Placebo

SUMMARY:
A double-blinded, placebo-controlled study of Dimethyl fumarate (DMF) in 34 Systemic Sclerosis-Pulmonary Hypertension (SSc-PAH) patients. The study will determine safety and the primary outcome variability for DMF in treating SSc-PAH; the primary outcome of clinical efficacy in this pilot trial will be improvement in 6-minute walk distance (6MWD).

DETAILED DESCRIPTION:
A double-blinded, placebo-controlled study of Dimethyl fumarate (DMF) in 34 Systemic Sclerosis-Pulmonary Hypertension (SSc-PAH) patients. The study medication will be added to stable background PAH medication(s). Subjects will be dosed for 24 weeks, will undergo examination every 8 weeks, and will be finally evaluated 12 weeks after completion of treatment. Dosage will begin at once daily oral doses of 120mg for the first 7 days and follow the up-titration schedule to a maintenance dose of 240mg twice a day (or highest tolerated dose of a minimum of 120mg twice a day by the start of Week 8) for the remainder of the study. Participation will be for a total of 40 weeks, including a 4-week screening period, 24 weeks of drug, and a safety follow-up 12 weeks after the last dose. The study will determine the safety and the primary outcome variability for DMF in treating SSc-PAH; the primary outcome of clinical efficacy in this pilot trial will be improvement in 6-minute walk distance (6MWD).

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent prior to any study-mandated procedures
2. Adult patients 18-80 years of age
3. World Health Organization Group 1 PAH associated with scleroderma (SSc-PAH)
4. WHO functional Class II-III
5. 6MWD 150 to 450 meters
6. Right heart catheterization demonstrating mPAP≥ 25 mmHg and PCWP or left ventricular end diastolic pressure ≤15mm Hg and pulmonary vascular resistance ≥240 dynes/cm-5 (3 Wood units) within 12 weeks prior to study entry.
7. ACR defined systemic sclerosis

Exclusion Criteria:

1. Pulmonary hypertension associated with

   * PAH of any etiology other than scleroderma
   * PH of any etiology other than WHO Group I PAH
   * Pulmonary venous hypertension defined as PCWP or LVEDP >15 mHg
   * Untreated sleep apnea with AHI >20 or SaO2 Nadir <87%
   * Chronic thromboembolic disease
   * Sarcoidosis
2. Participation in a clinical investigational study within the previous 30 days
3. Moderate to severe hepatic impairment (e.g., Child-Pugh Class B or C)
4. Renal failure defined as:

   * estimated creatinine clearance <30 m/min
   * serum creatinine>2.5 mg/dl
5. Serum aspartate aminotransferase (AST) and or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal
6. Systolic blood pressure < 90mmHg
7. Recently started (< 8 weeks prior to randomization) or planned cardiopulmonary rehabilitation program based on exercise
8. Pregnant or lactating women
9. Need for HAART therapy
10. Planned treatment or treatment with another investigational drug within 1 month prior to start
11. Moderate to severe interstitial lung disease, defined by FVC < 80% or evidence on HRCT of fibrosis or ground glass changes involving more than 30% of lung parenchyma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12; Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Lafyatis, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - National Jewish, Denver, Colorado
  - John Hopkins, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimethyl Fumarate (DMF): Once daily oral doses of Dimethyl Fumarate (DMF) 120mg for the first 7 days, following a titration schedule reaching a minimum of 120mg DMF twice daily, maximum 240mg twice daily, by the start of week 8. Subjects will be dosed for 24 weeks.
  Dimethyl Fumarate (DMF): Dimethyl Fumarate (DMF) is a prescription medicine used to treat relapsing multiple sclerosis.
Period: Overall Study
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Started | 4 | 2
Completed | 1 | 1
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Met stopping rule of low absolute lymphocyte count (<0.5L) at two visits | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dimethyl Fumarate (DMF) | Placebo | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Median (Full Range); unit: years] | 66.4 [45 to 71.7] | 72.5 [70.6 to 74.3] | 69 [45 to 74.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
6-minute walk distance (6MWD) [Mean (Full Range); unit: Mean 6MWD (meters)] | 305.5 [183 to 400] | 243.5 [183 to 304] | 284.83 [183 to 400]

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance (6MWD)
Description: The primary outcome of clinical efficacy in this study is improvement in 6-minute walk distance (6MWD). Data depict the mean change (%) at end-of-study-treatment (Week 24) from baseline in both treatment groups, utilizing the Last Observation Carried Forward of withdrawn subjects.
Time Frame: Baseline to Week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Number analyzed (Participants) | 4 | 2
percent change | -7.07 [-24.69 to 8.20] | -14.97 [-29.93 to 0]

2. Secondary Outcome: Clinical Worsening
Description: The change in time to clinical worsening in DMF compared to placebo treated patients.
Time Frame: Baseline to Week 24
Population: Insufficient data collection due to low recruitment and early termination of study.
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Borg Dyspnea Index (BDI)
Description: The change in Borg Dyspnea Index (BDI) at 24 weeks from baseline in DMF compared to placebo treated patients
Time Frame: Baseline to Week 24
Population: Insufficient data collection due to low recruitment and early termination of study.
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serum Markers of Oxidative Stress
Description: The change from baseline of serum markers of oxidative stress at 24 weeks, comparing DMF to placebo treated patients.
Time Frame: Baseline to Week 24
Population: Insufficient data collection due to low recruitment and early termination of study.
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proteomic Biomarkers
Description: The change from baseline in proteomic biomarkers, including BNP, at 24 weeks, comparing DMF to placebo treated patients.
Time Frame: Baseline to Week 24
Population: Insufficient data collection due to low recruitment and early termination of study.
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Dimethyl Fumarate (DMF) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (DMF) (N=4) | Placebo (N=2)
Worsening of heart failure and shortness of breath secondary to anemia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dimethyl Fumarate (DMF) (N=4) | Placebo (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Decreased CD4 lymphocytes (Investigations) | 1 (1) | 0 (0)
High cholesterol (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel bacteria overgrowth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Pneumonina (Infections and infestations) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Ankle swelling at night (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right rotator cuff tendinopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Early study termination due to low recruitment; not enough participants for statistically reliable analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT02981082/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02981082/ICF_001.pdf